CLINICAL TRIAL: NCT06881108
Title: Addressing Financial Hardship in Adolescent and Young Adult Cancer Survivors: Efficacy and Implementation of a Multilevel Intervention in Community-Based Oncology Practices
Brief Title: Addressing Financial Hardship in Adolescent and Young Adult Cancer Survivors
Acronym: FinFit Aim 1
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00107846; ONC-CCS-2410 (Other: Wake Forest Baptist Comprehensive Cancer Center); R01CA282653 (NIH); NCI-2025-01608 (Other: CTRP)
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Hematopoietic Neoplasm; Malignant Solid Neoplasm; Lymphatic System Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Observational step 1: CHAT participants complete an in-depth interview on study.
  Interventions: Other: CHAT Core Functions; Other: Member-Checking Process
- Observational step 2: LIFT participants complete a focus group or interview on study.
  Interventions: Other: LIFT Core Functions; Other: Member-Checking Process
- Observational step 3: Participants from steps 1 and 2 complete member-checking processes on study.
  Interventions: Other: Member-Checking Process

INTERVENTIONS:
Other: CHAT Core Functions — CHAT is a virtually delivered patient-level intervention designed to improve health insurance and cost-related literacy
  Groups: Observational step 1
Other: LIFT Core Functions — LIFT (Lessening the Impact of Financial Toxicity), an intervention developed to coordinate access to existing financial assistance programs.
  Groups: Observational step 2
Other: Member-Checking Process — Based on the findings from Steps 1 and 2, investigators will develop a document that outlines the points of overlap, harmony, or conflict identified by participants.

SUMMARY:
This study seeks to develop, test, and revise an intervention designed to address financial hardship (FinFit) among adolescent and young adult (AYA) cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To synthesize CHAT and LIFT to create FinFit, an intervention to address the unique, multilevel determinants of financial hardship among AYAs treated in community oncology practices.

OUTLINE: This is an observational study.

STEP 1: CHAT participants complete an in-depth interview on study.

STEP 2: LIFT participants complete a focus group or an interview on study.

STEP 3: Participants from steps 1 and 2 complete member-checking processes on study.

ELIGIBILITY:
Inclusion Criteria:

- Adults (ages 18 years of age or older) with perspectives on CHAT, LIFT, FinFit's proposed forms, and those from any community-based practices that were originally part of CHAT or LIFT administration are eligible for inclusion in Aim 1 interviews.

Exclusion Criteria:

- Those not involved in any of the preliminary programs, not familiar with the proposed forms of FinFit, or not involved in the proposed implementation sites will not be eligible for participation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with perspectives on CHAT, LIFT, and FinFit's proposed forms as well as individuals from any community-based practice that were originally part of CHAT or LIFT administration
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Combining Data Collection from Steps 1 and 2 for the Creation of FinFit Intervention Protocol | Up to 12 months
  Through the analysis of secondary outcomes (CHAT Core Functions - Step 1 LIFT Core Functions - Step 2) to develop, test, and revise an intervention designed to address financial hardship among adolescent and young adults using semi-structured interview data and analysis for the creation of protocol intervention including when, how and to whom the intervention should be delivered to.

SECONDARY OUTCOMES:
CHAT Core Functions - Step 1 | Up to 12 months
  Investigators will use ATLAS.ti, multifunctional qualitative data analysis software, to apply a codebook informed by the Model for Adaptation Design and Impact, and identify themes related to CHAT's core functions. Finally, we will use report-back sessions with interview participants to refine themes.
LIFT Core Functions - Step 2 | Up to 12 months
  Investigators will use ATLAS.ti, multifunctional qualitative data analysis software to apply grounded theory to analyze updates to existing LIFT core functions to apply a codebook informed by the Model for Adaptation Design and Impact, and identify themes related to CHAT's core functions and points of potential overlap, harmony, or conflict with LIFT's and CHAT's core functions using a 90-120 minute focus group to review previously identified core functions.
Member Checking Process - Step 3 | Up to 12 months
  Based on the findings from Steps 1 and 2, a document that outlines the points of overlap, harmony, or conflict identified by participants will be developed. Investigators will send this document back to all of the previous participants in a member-checking process, that will occur both virtually and asynchronously, to ensure the document reflects their perspectives. Once this document is finalized, investigators will draft the protocol for FinFit. Once drafted this document will be sent to all previous participants in a member-checking exercise for review and comment to ensure that it reflects their perspectives. The Model for Adaptation Design and Impact (MADI) tool will be used to evaluate potential points of overlap, harmony or conflict between the LIFT and CHAT steps to finally assess for potential influence on implementation outcomes (e.g. feasibility, acceptability) and FinFit outcomes (e.g., financial hardship).

CONTACTS AND LOCATIONS:
Overall Officials: John Salsman, PhD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No